CLINICAL TRIAL: NCT06913816
Title: Effects Of Optimized Blinking Training on Visual Function and Tear Film Parameters in Individuals With Computer Vision Syndrome
Brief Title: Effects Of Optimized Blinking Training on Visual Function and Tear Film Parameters in Individuals With CVS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall23/810
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Computer Vision Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grouyp 1 (without blinking exercises). (Active Comparator)
  Interventions: Diagnostic Test: Grouyp 1 (without blinking exercises).
- EXP group (Routine CVS treatment) (Experimental)
  Interventions: Combination Product: EXP group (Routine CVS treatment)

INTERVENTIONS:
Diagnostic Test: Grouyp 1 (without blinking exercises). — Group B (Control Group) The control group will continue receiving only the routine rehabilitation (without blinking exercises). Routine rehabilitation included the 20-20-20 rule, blue light-blocking glasses, and polyvinyl alcohol eye drops.
  Arms: Grouyp 1 (without blinking exercises).
Combination Product: EXP group (Routine CVS treatment) — "Group A (Experimental Group): Individuals in the Experimental group will receive Routine CVS treatment with optimized blinking exercise.
  Routine rehabilitation includes the 20-20-20 rule, blue light-blocking glasses, and polyvinyl eye drops.
  The blinking exercise involved the individuals looking at an object 6 meters away for 5 seconds, followed by complete eyelid closure for 5 seconds. This cycle was repeated for 5 minutes, twice a day."
  Arms: EXP group (Routine CVS treatment)

SUMMARY:
"Computer vision syndrome (CVS), refers to a range of eye and vision issues caused by extended use of computers, tablets, e-readers, and smartphones. Computer users experience visual symptoms, such as eyestrain, headaches, eye discomfort, dry eyes, double vision, and blurred vision, especially after long periods of looking at screens, whether up close or at a distance.

DETAILED DESCRIPTION:
Individuals will be randomly assigned to either an experimental group (group A) receiving OBT with routine rehabilitation CVS management 20-20-20 rule, blue light-blocking glasses, and polyvinyl alcohol eye drops or a control group (group B) receiving only routine rehabilitation, including the 20-20-20 rule, blue light-blocking glasses, and polyvinyl alcohol eye drops. OBT consisted of structured blinking exercises performed thrice daily for three months. Objective outcomes, including tear film parameters and visual function using subjective Computer Vision Syndrome Questionnaire (CVS-Q) shall be evaluated. The collected data will be analysed by using SPSS."

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-40 years who work on computers or digital devices for at least 3 to 6 hours daily.
* Both Male and Female.
* Individuals who could undergo a complete ocular examination.
* Presence of symptoms consistent with digital eye strain.
* Presented with eye complaints such as eye fatigue, burning, irritation, redness, and blurred vision due to long-term computer or digital screen use.
* Symptoms worsened during exposure to digital screen light.

Exclusion Criteria:

* Use of medications that might influence tear production or ocular surface status (e.g., antihistamines, antidepressants).
* Diagnosed neurological or systemic conditions that impact vision or blink patterns (e.g., Parkinson's disease, multiple sclerosis).
* Individual's with a history of ocular surface diseases such as conjunctivitis or keratitis.
* History of any psychiatric diagnosis."

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Computer Vision Syndrome (CVS-Q) | 12 Months
  The Computer Vision Syndrome Questionnaire (CVS-Q) assesses the frequency and intensity of 16 ocular and visual symptoms related to prolonged screen use, with a total score of 6 or more indicating CVS If the total score is ≥6 points, the individual is considered to suffer Computer Vision Syndrome

CONTACTS AND LOCATIONS:
Locations (1):
- Ramzan Eye Care and Optix Khudian Khas, Kasur, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No